CLINICAL TRIAL: NCT04674345
Title: Sorafenib Maintenance for Prophylaxis of Leukemia Relapse in Allogeneic Hematopoietic Stem Cell Transplant Recipients With FLT3 Negative Acute Leukemia
Brief Title: Sorafenib Maintenance for Prophylaxis of Leukemia Relapse in Allo-HSCT Recipients With FLT3 Negative Acute Leukemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Xiangya Hospital of Central South University (Other); Zhujiang Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); First People's Hospital of Chenzhou (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); The Third Xiangya Hospital of Central South University (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sorafenib-Non-Flt3 AL-2020
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2020-12

CONDITIONS: Acute Leukemia; Relapse; Hematopoietic Stem Cell Transplantation
Keywords: Acute Leukemia; Sorafenib; Relapse; FLT3-negative; Allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Recurrence | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sorafenib group (Experimental): Sorafenib will be administered at 45-60 days post-transplantation and taken for one year.
  Interventions: Drug: Sorafenib
- Non-maintenance group (No Intervention): Neither sorafenib nor other FLT3 inhibitors will be used, unless the patient experiences relapse.

INTERVENTIONS:
Drug: Sorafenib — The initial dose of sorafenib is 400 mg orally twice daily and is adjusted in case of suspected toxicity (dose range, 200-800 mg daily).
  Arms: Sorafenib group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of sorafenib maintenance after allo-HSCT in FLT3-negative acute leukemia patients.

DETAILED DESCRIPTION:
Sorafenib is a multikinase inhibitor that blocks multiple pathways involved in the development and progression of acute leukemia, such as FLT3-ITD, the RAS and RAF gene families, KIT, and the VEGF and PDGF receptors. Recently, two back-to-back randomized controlled trials both reveal that sorafenib maintenance after allo-HSCT could prevent relapse in patients with FLT3-ITD AML, resulting in a survival benefit. Sorafenib has also been explored in the treatment of acute leukemia without FLT3 mutations and shown promising results. Currently, relapse remains the major cause of transplant failure, especially for high-risk and refractory acute leukemia patients. Once patients relapse after allo-HSCT, the prognosis is dismal. Therefore, prevention of relapse is of great importance to improve the prognosis. Based on the current research status, we plan to conduct a prospective, multicenter, phase 2 randomized controlled trial to explore the efficacy and safety of sorafenib maintenance after allo-HSCT in FLT3-negative acute leukemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FLT3-negative acute leukemia undergoing first allo-HSCT
* Age 18 to 65 years old with ECOG performance status 0-2
* Hematopoietic recovery within 60 days post-transplantation
* Sign informed consent form, have the ability to comply with study and follow-up procedures

Exclusion Criteria:

* Acute promyelocytic leukemia (AML subtype M3)
* Acute leukemia with FLT3-ITD or FLT3-TKD mutations
* Philadelphia-positive acute lymphoblastic leukemia
* Chronic myelogenous leukemia with blast crisis
* Intolerance to sorafenib pre-transplantation
* Life expectancy less than 30 days post-transplantation
* Active aGVHD or uncontrolled infections within 60 days post-transplantation
* Cardiac dysfunction (particularly congestive heart failure, unstable coronary artery disease and serious cardiac ventricular arrhythmias requiring antiarrhythmic therapy)
* Respiratory failure ( PaO2 ≤60mmHg)
* Hepatic abnormalities (total bilirubin ≥3 mg/dL, aminotransferase >2 times the upper limit of normal)
* Renal dysfunction (creatinine clearance rate < 30 mL/min)
* ECOG performance status 3, 4 or 5
* With any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of leukemia relapse | 1 year

SECONDARY OUTCOMES:
Overall survival | 1 year
Leukemia-free survival | 1 year
Adverse effects | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China